CLINICAL TRIAL: NCT04400656
Title: PROState Pathway Embedded Comparative Trial
Acronym: IP3-PROSPECT
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Imperial Clinical Trials Unit (ICTU) (Unknown); Wellcome Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 19CX5601
Record Dates: First submitted 2020-05-11; First posted 2020-05-22 (Actual); Results first posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer; Non-metastatic Prostate Cancer; Metastatic Prostate Cancer; Prostate Adenocarcinoma; Metastatic Prostate Carcinoma in the Soft Tissue; Prostate Cancer Metastatic
Keywords: prostate cancer; Non-metastatic Prostate Cancer; Metastatic Prostate Cancer; Prostate Adenocarcinoma; Metastatic Prostate Carcinoma in the Soft Tissue; Prostate Cancer Metastatic; Clinical Trial Design; cohort multiple randomised controlled trial; cmRCT; Trials Within Cohorts; TWICS
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The proposal will explore a trial design called the cohort-multiple RCT (cmRCT) or as it has been recently coined, the Trials WithIn Cohorts (TWICS) design. This design has been used in a number of disease areas, both benign and cancer. Prostate conditions have been chosen since they are extremely common and if malignancy occurs the majority of men with the disease are regarded as living with a chronic condition due to its long natural history and in which innovative approaches, interventions, treatments or changes in management might have a significant patient benefit and impact on the NHS. It therefore fits the cmRCT design very well. Nonetheless, the lessons learned in this study will be of relevance to other disease spaces.

The TWICS or cmRCT design is currently being used in elderly patients, risk of falls, depression, hip fracture, Yorkshire Health Study, scleroderma, breast cancer, colorectal cancer, bladder cancer and kidney cancer, to name a few. In total, a recent systematic review showed that there were 18 ongoing cmRCT studies with 6 in the UK.

The acceptability and feasibility of the cmRCT in the prostate pathway will be tested. This is the first time this method will be tested and therefore piloted. In the first part of the study, the following will be evaluated. What is the accrual rate? What do patients and their healthcare professionals think of the cmRCT design? Is the data collected robust? What are the resource requirements of such a study?A number of novel interventions or changes in the pathway will then be tested and compared to standard care in the cohort that was recruited.

DETAILED DESCRIPTION:
TRIAL AIMS

The pilot phase of PROSPECT is interested in investigating the a) acceptability and feasibility of establishing the cohort of men, i.e. putting the questions of Point of Consent One to men being referred for investigation of prostate cancer, and b) observing the cohort over the study period and collecting data on the participants pertaining to their disease, their treatment and their health status.

A) Acceptability

AIM 1.1: To determine what proportion of men with a clinical suspicion for prostate cancer will participate in an cmRCT.

OBJECTIVE 1.1a: To evaluate proportion of patients approached who agree to participate in the longitudinal cohort. This will be done by calculating the participation rates from men approached for invitation to PROSPECT.

AIM 1.2: To explore barriers and facilitators to implementation of a cmRCT in order to improve and inform patient and/or physician trial information, study processes, interventions, and recruitment and retention of patients. This will be carried out by qualitative assessments in the following areas.

OBJECTIVE 1.2a: To investigate by interview the patient experiences and perspectives on;

* Trial participation,
* The point at which men are approached by the research team to enter the cohort,
* Barriers and facilitators to consent to participate in the cohort,
* Barriers and facilitators to consent to future random selection to undergo a new healthcare intervention,
* Acceptability of monitoring of health status and the tools used to do this in the cohort.

OBJECTIVE 1.2b: To investigate by interview the experiences and perspectives of healthcare professionals (doctors, nurses and admin staff) on;

* Trial design and information to patients and healthcare professionals,
* Feasibility of future random invitation of participants to interventions,
* Tools used for measuring health status.

B) FEASIBILITY

AIM 2.1: To determine the feasibility of recruitment and logistical implementation of PROSPECT in different data collecting centres based in different institutions. This will be broken down into the following sub-questions;

OBJECTIVE 2.1a: Evaluating how the patients are successfully identified and the option of how inclusion in the trial is presented to them.

OBJECTIVE 2.1b: Evaluate patient questionnaire response rates for pre-treatment quality of life.

OBJECTIVE 2.1c: Evaluate patient questionnaire response rates at pre-determined intervals following on from the point of recruitment into the trial to determine how to promote optimal patient response rate and improve data collection.

OBJECTIVE 2.1d: To evaluate completeness and fidelity of clinical data on the men who participate in the cohort.

STUDY DESIGN

Design

The key features of a cmRCT are;

1. Explicitly consented recruitment of a large cohort of patients with the condition of interest.
2. Regular measurement of relevant outcome measures for the whole cohort prospectively in the long-term.
3. Facility to re-approach cohort participants, who are randomly selected from eligible patients within the cohort, inviting them to undergo intervention of interest to researchers with eligible patients not randomly selected entering the control standard care group (see study flowchart 3.3 / 3.4).
4. "Patient-centred" informed consent. The consent process aims to replicate that used in the routine health care setting. Once the patient has been randomly selected for a randomised novel intervention from the eligible patients within the cohort, the second consent process should include detailed and specific information pertaining to the particular intervention or change in management they are being invited to undergo for comparison. Such information will be written and advised using patient representatives and undergo review following submission to REC.
5. Comparison of the outcomes in the randomly selected patients with the outcomes in eligible patients not randomly selected.
6. Capacity for multiple randomised controlled trials over time within the cohort simultaneously.

CONSENT

For men who are participating in the cmRCT there are two points of consent:

POINT OF CONSENT ONE

At Point of Consent One men who are referred for investigation of prostate cancer will be asked two questions. The first question relates to whether they are willing to join the cohort and have data collected directly from them over time on a regular basis. This data will include health-related quality-of-life data (at recruitment, 0-6, 6, 12, 18 & 24 months post recruitment), linkage to their medical records so that researchers can know what happens to them over time, and access to other data about them held on national health registry databases. Also, at point of consent one, prospective participants will be asked (second question) whether they agree to being randomly selected in the future to interventions or changes in management in order to compare to standard care. It will be explained that this second invitation will be on a random basis. In other words, everyone eligible within the cohort will have the same chance of being randomly selected. The patient would still have the option of saying 'no' after the random selection when they are approached.

POINT OF CONSENT TWO

The second point of consent is the invitation to undergo an intervention or change in management that the research team wishes to compare to standard care. Participants will have already agreed to the possibility of being invited to undergo intervention at Point of Consent One (i.e. enrolment into the cmRCT). The participant will have been randomly selected from amongst all the eligible men for the given intervention from within the large cmRCT cohort prior to being approached by the trial team. Then, the trial team will approach the participant and invite him to undergo the intervention. This will entail a comprehensive consent process that pertains directly to the intervention being proposed in a patient-centred manner. The participant can agree or refuse to undergo the intervention. If he does not wish to undergo the treatment he will continue under follow-up in PROSPECT.

Participants undergoing intervention will continue to have follow-up in the same manner as men who have not been randomised from within the cohort and thus provide outcome data to form the control arm. Comparison of the outcomes of those men who underwent trial intervention against those who did not will allow us to analyse the effectiveness of the intervention in as robust a manner as possible given that the key feature of randomisation when creating the control vs. the intervention arms has been preserved. As such, the control arm of the cmRCT will be similar to the intervention arm in all features, known and unknown, except the intervention of interest. This will allow for the maintenance of epistemological superiority of the data produced for evaluating new tests or treatments whilst getting to this point in a way that might be more acceptable to patients and therefore more likely to be successful and efficient for researchers.

The second stage of PROSPECT will be to investigate and evaluate in a similarly careful manner the feasibility and acceptability of randomising men from the cohort of eligible men to interventions or changes in management that require evaluation, following submission to REC. As part of the cmRCT design, these men randomly selected are re-approached and invited to consider undergoing the intervention of interest. Patients who are randomly allocated to the control arm will also receive standard of care, and are not informed about their participation in the control arm. This additional consent will be obtained at the time of consent for the cohort study.

STUDY SETTING AND POPULATION

All men referred for investigation of prostate cancer. The inclusion criteria for this cohort is deliberately broad.

ELIGIBILITY:
Inclusion Criteria:

1. Men aged 18 years old and over who are referred for investigations for urinary symptoms or elevated serum prostate specific antigen (PSA) levels or other risk factors for possible prostate malignancy.
2. An understanding of the English language sufficient to understand written and verbal information about the trial and consent process.
3. Estimated life expectancy of 5 years or more.
4. Signed informed consent.

Exclusion Criteria:

1. Men who are unable to give informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men with possible prostate malignancy
Study Population: All men referred for investigation of prostate cancer
Sampling Method: Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hashim Ahmed, Principal Investigator — Imperial College London
Locations (3):
- United Kingdom (3):
  - West Middlesex University Hospital, Isleworth, Middlesex
  - Ashford & St Peter's Hospitals (ASPH) NHS Foundation Trust, Chertsey, Surrey
  - Imperial College Healthcare NHS Trust, London

REFERENCES:
- [Derived] Peters M, Eldred-Evans D, Kurver P, Falagario UG, Connor MJ, Shah TT, Verhoeff JJC, Taimen P, Aronen HJ, Knaapila J, Montoya Perez I, Ettala O, Stabile A, Gandaglia G, Fossati N, Martini A, Cucchiara V, Briganti A, Lantz A, Picker W, Haug ES, Nordstrom T, Tanaka MB, Reddy D, Bass E, van Rossum PSN, Wong K, Tam H, Winkler M, Gordon S, Qazi H, Bostrom PJ, Jambor I, Ahmed HU. Predicting the Need for Biopsy to Detect Clinically Significant Prostate Cancer in Patients with a Magnetic Resonance Imaging-detected Prostate Imaging Reporting and Data System/Likert >/=3 Lesion: Development and Multinational External Validation of the Imperial Rapid Access to Prostate Imaging and Diagnosis Risk Score. Eur Urol. 2022 Nov;82(5):559-568. doi: 10.1016/j.eururo.2022.07.022. Epub 2022 Aug 11. PMID 35963650

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Acceptability and Feasibility sample size: 80 patients. However the actual cohort sample will not be restricted as the overall number needed will be dependent on future randomised interventions and therefore there is no maximum number. If the feasibility number is met then we will continue recruiting for the entire recruitment period with no upper limit on numbers and continue beyond the existing recruitment period if further funding allows and pending approval by REC.
Groups:
- Acceptability and Feasibility Group: Men who have been referred for further investigation due to elevated PSA, lower urinary tract symptoms or abnormal rectal examinations
Period: Overall Study
Arm/Group | Acceptability and Feasibility Group
Started | 139
Completed | 139
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Feasibility Group - Age, Ethnicity, BMI, PSA DRE & WHO Performance Status: Feasibility Group- patients referred for prostate investigations.
  Age, Ethnicity, BMI, PSA DRE & WHO Performance Status
Arm/Group | Feasibility Group - Age, Ethnicity, BMI, PSA DRE & WHO Performance Status
Number analyzed (Participants) | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 139
Race/Ethnicity, Customized [Number; unit: participants]
  White | 116
  Mixed / Multiple Ethnic Groups | 2
  Asian / Asian British | 7
  Black / African / Caribbean / Black British | 4
  Other Ethnic Group | 5
  Unknown | 5
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body mass index (BMI) is a measure of body fat based on height and weight Population: 37 entries missing from eCRF
  kg/m^2
    number analyzed (Participants) | 102
    (all) | 26.31 (5.14)
PSA [Mean (Standard Deviation); unit: ng/mL] — A blood test taken to determine the level of Prostate-specific antigen (PSA) in nanograms per milliliter within the blood Population: 1 entry missing from eCRF
  ng/mL
    number analyzed (Participants) | 138
    (all) | 6.41 (3.28)
DRE [Number; unit: participants] — Digital rectal examination (DRE), also known as a prostate exam is an internal examination of the rectum performed by a healthcare provider. Population: 10 entries missing from eCRF
  participants
    No: number analyzed (Participants) | 129
    No | 96
    Yes- (but DRE result missing): number analyzed (Participants) | 129
    Yes- (but DRE result missing) | 1
    Yes-Abnormal: number analyzed (Participants) | 129
    Yes-Abnormal | 7
    Yes-Evidence for Locally Advanced/Metastatic Disease: number analyzed (Participants) | 129
    Yes-Evidence for Locally Advanced/Metastatic Disease | 1
    Yes-Normal: number analyzed (Participants) | 129
    Yes-Normal | 24
WHO Performance Status [Number; unit: participants] — The healthcare providers grading of a patient based on The World health Organisation (WHO) performance status classification from the below:
  0: able to carry out all normal activity without restriction
  1. restricted in strenuous activity but ambulatory and able to carry out light work
  2. ambulatory and capable of all self-care but unable to carry out any work activities; up and about more than 50% of waking hours Population: 1 entry missing from the eCRF
  participants
    0: number analyzed (Participants) | 138
    0 | 125
    1: number analyzed (Participants) | 138
    1 | 10
    2: number analyzed (Participants) | 138
    2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Men Who Consented to Inclusion in PROSPECT Study Out of Total Number of Patients Approached
Description: Number of men who consented to inclusion in PROSPECT Study out of total number of patients approached at the original point of contact by the research team.
Time Frame: from baseline to 23 months
Population: Number analysed in the approached rate refers to the number of patients reffered to the study but may not have joined the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Acceptability Endpoint - Consent Rate: Proportion of patients who consented to inclusion in PROSPECT cohort out of total number of patients approached
Arm/Group | Acceptability Endpoint - Consent Rate
Number analyzed (Participants) | 384
percentage of participants | 36.2 [31.4 to 41.2]

2. Primary Outcome: Number of Participants Approached for the Study From the Number of Patients Referred to the Study Team by Other Participating Centres
Description: Evaluation of the number of men approached to enter the PROSPECT Study from the number of men referred to the participating centres for investigation of prostate cancer.
Time Frame: from baseline to 23 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Acceptability Endpoint - Approached Rate: Proportion of men approached to enter PROSPECT out of number of men referred to the participating centres for investigation of prostate cancer
Arm/Group | Acceptability Endpoint - Approached Rate
Number analyzed (Participants) | 462
percentage of participants | 83.1 [79.4 to 86.4]

3. Primary Outcome: Number of Participants Who Complete a Questionnaire on the Quality of Life (EQ5D-5L)
Description: Number of Participants who complete a given standard Quality of Life Questionnaire (EQ5D-5L) at the point at which they consent to inclusion into PROSPECT. (Baseline Visit)
Time Frame: Questionnaire was completed at baseline - 0 months, visit 1 - 6 months, visit 2 -12 months and visit 3 -18 months.
Population: Number of patients who responded/started the questionnaire & number of patients who completed the questionnaire
Measure: Count of Participants; unit: Participants
Groups:
- Completeness of EQ5D-5L Data - Proportion Responded; Completeness of EQ5D-5L Data - Proportion Completed: Participants will be given a standard Quality of Life Questionnaire (EQ5D-5L) at the point at which they consent to inclusion into PROSPECT. We will calculate the completeness of this data one year after opening and on an ongoing basis.
Arm/Group | Completeness of EQ5D-5L Data - Proportion Responded | Completeness of EQ5D-5L Data - Proportion Completed
Number analyzed (Participants) | 139 | 139
Participants
  Visit 0 (Baseline) | 109 | 109
  Visit 1 (6 months) | 96 | 96
  Visit 2 (12 months) | 95 | 93
  Visit 3 (18 months) | 24 | 24

4. Primary Outcome: Number of Participants Who Complete a Questionnaire on Quality of Life (EPIC-26)
Description: Number of Participants who completed a given standard Quality of Life Questionnaire (EPIC-26) at the point at which they consent to inclusion into PROSPECT. (Baseline Visit)
Time Frame: Questionnaire was completed at baseline - 0 months, visit 1 - 6 months, visit 2 -12 months and visit 3 -18 months.
Population: Number of patients who responded/started the questionnaire & number of patients who completed the questionnaire
Measure: Count of Participants; unit: Participants
Groups:
- Completeness of EPIC-26 Data - Proportion Responded; Completeness of EPIC-26 Data - Proportion Completed: Participants will be given a standard Quality of Life Questionnaire (EPIC-26) at the point at which they consent to inclusion into PROSPECT. We will calculate the completeness of this data one year after opening and on an ongoing basis.
Arm/Group | Completeness of EPIC-26 Data - Proportion Responded | Completeness of EPIC-26 Data - Proportion Completed
Number analyzed (Participants) | 139 | 139
Participants
  Visit 0 (Baseline) | 110 | 107
  Visit 1 (6 months) | 96 | 96
  Visit 2 (12 months) | 93 | 87
  Visit 3 (18 months) | 24 | 22

5. Primary Outcome: Number of Participants Who Complete a Questionnaire on Quality of Life (IPSS)
Description: Number of Participants who complete a given standard Quality of Life Questionnaire (IPSS) at the point at which they consent to inclusion into PROSPECT.
Time Frame: Questionnaire was completed at baseline - 0 months, visit 1 - 6 months, visit 2 -12 months and visit 3 -18 months.
Population: Number of patients who responded/started the questionnaire & number of patients who completed the questionnaire
Measure: Count of Participants; unit: Participants
Groups:
- Completeness of IPSS Data - Proportion Responded; Completeness of IPSS Data - Proportion Completed: Participants will be given a standard Quality of Life Questionnaire (IPSS) at the point at which they consent to inclusion into PROSPECT. We will calculate the completeness of this data one year after opening and on an ongoing basis.
Arm/Group | Completeness of IPSS Data - Proportion Responded | Completeness of IPSS Data - Proportion Completed
Number analyzed (Participants) | 139 | 139
Participants
  Visit 0 (Baseline) | 109 | 107
  Visit 1 (6 months) | 97 | 96
  Visit 2 (12 months) | 93 | 92
  Visit 3 (18 months) | 24 | 23

6. Primary Outcome: Number of Participants Who Complete a Questionnaire on Quality of Life (IIEF-15)
Description: Number of Participants who completed a given standard Quality of Life Questionnaire (IIEF-15) at the point at which they consent to inclusion into PROSPECT. (Baseline Visit)
Time Frame: Questionnaire was completed at baseline - 0 months, visit 1 - 6 months, visit 2 -12 months and visit 3 -18 months.
Population: Number of patients who responded/started the questionnaire & number of patients who completed the questionnaire
Measure: Count of Participants; unit: Participants
Groups:
- Completeness of IIEF-15 Data - Proportion Responded: Participants will be given a standard Quality of Life Questionnaire (IPSS) at the point at which they consent to inclusion into PROSPECT. We will calculate the completeness of this data one year after opening and on an ongoing basis.
- Completeness of IIEF-15 Data - Proportion Completed: Participants will be given a standard Quality of Life Questionnaire (IIEF-15) at the point at which they consent to inclusion into PROSPECT. We will calculate the completeness of this data one year after opening and on an ongoing basis.
Arm/Group | Completeness of IIEF-15 Data - Proportion Responded | Completeness of IIEF-15 Data - Proportion Completed
Number analyzed (Participants) | 139 | 139
Participants
  Visit 0 (Baseline) | 107 | 99
  Visit 1 (6 months) | 96 | 88
  Visit 2 (12 months) | 91 | 86
  Visit 3 (18 months) | 23 | 20

ADVERSE EVENTS:
Time Frame: 23 months
Description: An AE is any untoward medical occurrence in a patient or clinical trial subject. For the purposes of the study, all AEs and SAEs were recorded throughout the study, however none are associated with the study itself as PROSPECT is an observational study only.
Groups:
- Summary of Adverse Events: Summary of Adverse events from Feasibility Group
Arm/Group | Summary of Adverse Events
All-Cause Mortality (participants affected / at risk) | 0/139
Serious Adverse Events (participants affected / at risk) | 3/139
Other Adverse Events (participants affected / at risk) | 78/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Summary of Adverse Events (N=139)
Incision and drainage, hospital admission (Surgical and medical procedures) | 1 (1)
Left Ring Finger fracture (Injury, poisoning and procedural complications) | 1 (1)
Psychosis (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Summary of Adverse Events (N=139)
Abnormal gait (General disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Ataxia (General disorders) | 1 (1)
Back pain (General disorders) | 2 (2)
COVID 19 infection (Infections and infestations) | 2 (2)
Catheter pain (Renal and urinary disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cognitive dysfunction (Psychiatric disorders) | 1 (1)
Community acquired pneumonia (Immune system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diarrhoea and vomiting (Gastrointestinal disorders) | 1 (1)
Erectile Dysfunction (Renal and urinary disorders) | 7 (7)
Faecal Frequency (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Flare of ulcerative Colitis (Gastrointestinal disorders) | 1 (1)
Groin abscess (Skin and subcutaneous tissue disorders) | 1 (1)
Haematospermia (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2)
Head injury (General disorders) | 1 (1)
Headaches (General disorders) | 1 (1)
High post void residual volumes (Renal and urinary disorders) | 1 (1)
Hip sprain (Injury, poisoning and procedural complications) | 1 (1)
Hot flashes (General disorders) | 3 (3)
Inguinal Hernia repair (Surgical and medical procedures) | 1 (1)
Intermittent Confusion (Psychiatric disorders) | 1 (1)
Knee pain (General disorders) | 1 (1)
Left Ring Finger fracture (Injury, poisoning and procedural complications) | 1 (1)
Leg pain (General disorders) | 1 (1)
Loss of balance (General disorders) | 1 (1)
Low urinary flow rate (Renal and urinary disorders) | 1 (1)
Lower urinary tract symptoms (Renal and urinary disorders) | 6 (6)
Nocturia (Renal and urinary disorders) | 2 (2)
Perineal pain (Renal and urinary disorders) | 1 (1)
Poor urinary flow (Renal and urinary disorders) | 1 (1)
Post traumatic epilepsy (Psychiatric disorders) | 1 (1)
Post traumatic stress disorder (Psychiatric disorders) | 1 (1)
Prostatitis (Infections and infestations) | 1 (1)
Psychosis (Psychiatric disorders) | 1 (1)
Pyelonephritis (Renal and urinary disorders) | 1 (1)
Recurrent Urinary Tract Infections (Renal and urinary disorders) | 2 (2)
Reduced ejaculatory volume (Renal and urinary disorders) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1)
Right groin pain (General disorders) | 1 (1)
Sprained ankle (Injury, poisoning and procedural complications) | 1 (1)
Stress Urinary Incontinence (Renal and urinary disorders) | 1 (1)
Total hip arthroplasty (Surgical and medical procedures) | 1 (1)
Transient Ischaemic Attack (Vascular disorders) | 1 (1)
Tremor (Musculoskeletal and connective tissue disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 2 (2)
Watery stool (Gastrointestinal disorders) | 1 (1)
Weight gain (General disorders) | 1 (1)
Worsening shortness of breath (General disorders) | 1 (1)
calf swelling (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-04-05): https://cdn.clinicaltrials.gov/large-docs/56/NCT04400656/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/56/NCT04400656/SAP_001.pdf